CLINICAL TRIAL: NCT05397002
Title: Patient Specific Intraoral Inverted-L Osteotomy Modified With Inferior Alveolar Nerve Relocation in Corrective Mandibular Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohammed Abdel Salam Ibrahim Omara, Lecturer, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OMFS -1-10-20
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Class III Malocclusion
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with class III malocclusion (Other)
  Interventions: Procedure: patient specific inverted L mandibular osteotomy modified with inferior alveolar nerve relocation

INTERVENTIONS:
Procedure: patient specific inverted L mandibular osteotomy modified with inferior alveolar nerve relocation — preoperative CBCT was requested for virtual planning and fabrication of cutting and drilling guides. Cutting lines were outlined to be consisted of four cuts; lateral ostectomy to uncover and lateralize the inferior alveolar nerve (IAN), posterior cut run horizontally from the anterior border of the ramus to a point just above the mandibular foramen, two anterior vertical cuts run from the anterior end of the lateral ostectomy to the inferior mandibular border. The guide was removed and the osteotomy lines were completed then the mandibular setback was oriented and fixed using pre-bent plates osteosynthesis. Plane transfer was checked using CBCT and Inferior alveolar nerve function was assessed.

SUMMARY:
Bilateral sagittal split osteotomy (BSSO) is considered the main osteotomy design in corrective mandibular surgery, however abnormal anatomical configuration of the posterior mandible with rolled out inferior border and thin mandibular rami with cortically adherent inferior alveolar nerve may interfere with the utilization of this osteotomy. The aim of this study is to introduce a novel modification of the intraoral inverted L ramus osteotomy (ILRO) to overcome these limitations in mandibular setback surgery. preoperative CBCT was requested for virtual planning and fabrication of cutting and drilling guides. Cutting lines were outlined to be consisted of four cuts; lateral ostectomy to uncover and lateralize the inferior alveolar nerve (IAN), posterior cut run horizontally from the anterior border of the ramus to a point just above the mandibular foramen, two anterior vertical cuts run from the anterior end of the lateral ostectomy to the inferior mandibular border. The guide was removed and the osteotomy lines were completed then the mandibular setback was oriented and fixed using pre-bent plates osteosynthesis. Inferior alveolar nerve function was regained perfectly one year post-operatively. This procedure introduces a robust alternative to the BSSO osteotomy in some cases of mandibular setback surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients.
* patients with skeletal class III malocclusion.
* Patients with thin mandibular rami with minimal medullary bone.
* Patients with inferior alveolar nerve proximity to the buccal cortex.
* Patients with lateral bending of the inferior mandibular border at molar angle region.
* Patients with high mandibular foramen.

Exclusion Criteria:

* Patients with previous extensive jaw surgery.
* mandibular pathological lesions.
* Patients with temporomandibular joint dysfunction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-04-10 (Actual); Study Completion 2022-04-10 (Actual)

PRIMARY OUTCOMES:
Neurosensory dysfunction of Inferior Alveolar Nerve | one year after surgical intervention
  Neurosensory test: two-point discrimination test

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Omara, Lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No